CLINICAL TRIAL: NCT01740037
Title: IntegRAted Chronic Care Program at a Specialized Atrial Fibrillation (AF) Clinic Versus Usual CarE in Patients With Atrial Fibrillation, an Investigator-initiated, Prospective, Randomised, Open Label, Blinded Outcome Assessment (PROBE) Controlled Multi-center Study
Brief Title: IntegRAted Chronic Care Program at Specialized AF Clinic Versus Usual CarE in Patients With Atrial Fibrillation - RACE4
Acronym: RACE4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Stichting Achmea Gezondheidszor (Other); DSW (Unknown); CZ Fonds (Other); Bayer (Industry); Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry); Pfizer (Industry); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METC 11-2-099
Record Dates: First submitted 2012-10-16; First posted 2012-12-04 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
Keywords: Integrated chronic care program; specialized outpatient AF clinic; Atrial Fibrillation guideline
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Specialized AF-clinic (Experimental): Management of AF patients in specialized outpatient AF Clinics according to the principles of an integrated chronic care program (ICCP) performed by a nurse practitioner/ physician assistant/ specialised cardiovascular nurse, cardiologist, supported by an ICT decision support tool based on professional guidelines (CardioConsult AF®). The use of a web-based patient centered management of patient's own medication (Medication manager TM) was optional. A standardized diagnostic, treatment and follow-up pathway was performed within the ICCP. In addition, the intervention is based on identifying risk factors and potential problems in patients, and addressing needs through dynamic use of personalized education and adjustment of treatment.
  Interventions: Other: Specialized outpatient AF Clinic
- Usual Care (Active Comparator): Usual care provided by cardiologists at the regular outpatient clinic.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Specialized outpatient AF Clinic
  Arms: Specialized AF-clinic
Other: Usual Care
  Arms: Usual Care

SUMMARY:
Rationale: The treatment of patients with atrial fibrillation is often inadequate due to poor guideline adherence. An integrated chronic care program (ICCP) at a specialized AF-clinic was found to be superior to usual care provided by a cardiologist in terms of cardiovascular hospitalizations and cardiovascular mortality.

Hypothesis: treatment at a specialized AF clinic is superior to usual care in terms of cardiovascular mortality and cardiovascular hospitalizations, cost-effectiveness, quality of life and guideline adherence.

Objectives: primary objective is to show that an ICCP reduces cardiovascular hospitalizations and mortality.

Study design: randomized controlled trial with two study arms: usual care provided by cardiologists (control) versus integrated chronic care program at a specialized AF clinic (intervention) in 8 hospitals in the Netherlands. The RACE4 is an event driven study. A total number of 246 events is needed. In total 1716 patients with newly diagnosed AF will be included. Total duration of the study is 5 years and 10 months with a minimal follow up of 1 year. Data is collected at inclusion, after 3, 6, 12 months, every year thereafter and at the end of the study.

Study population: Patients older than 18 year with newly diagnosed AF.

Intervention: The intervention is delivered through the specialized outpatient AF clinic. The multidisciplinary team at the AF clinic consists of a nurse practitioner or physician assistant or specialised cardiovascular nurse, cardiologist, and is guided by guidelines-based decision support software program based on the applicable ESC guideline recommendations. The use of a web-based patient centered management of patient's own medication (Medication manager TM) was optional. A standardized diagnostic, treatment and follow-up pathway was performed within the ICCP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed AF detected on electrocardiogram (ECG), holter recordings or event recorder with a duration > 30 seconds, 3 months before inclusion or
2. Patients with a history of diagnosed AF, with no regular control at a cardiologist for AF in the last 2 years and referred by a (non-)cardiologic medical specialist for new diagnostics or therapeutic issue;
3. Age ≥18 years.

Exclusion Criteria:

1. No electrocardiographic objectified AF;
2. Unstable heart failure defined as NYHA IV or heart failure necessitating hospital admission < 3 months before inclusion;
3. Acute coronary syndrome (acute myocardial infarction or instable angina pectoris, with two of the following characteristics: chest pain and/ or ischemic electrocardiographic changes, and/ or cardiac enzyme rise) < 3 months before inclusion;
4. Untreated hyperthyroidism or < 3 months euthyroidism before inclusion;
5. Foreseen pacemaker, internal cardioverter defibrillator, and/ or cardiac resynchronization therapy;
6. Cardiac surgery ≤ 3 months before inclusion;
7. Planned cardiac surgery;
8. Regular control and treatment, also for AF, at another specialized outpatient cardiac clinic;
9. Patient is not able to fill in the questionnaires;
10. Participation in other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1375 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a composite of unplanned admission to the hospital for any cardiovascular reason and cardiovascular death. | Follow up with minimum of 1 year and a maximum of 5 years and 10 months

SECONDARY OUTCOMES:
All components of the primary endpoint | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
All-cause mortality | Minimum of 1 year and a maximum of 5 years and 10 months
Total number of unplanned all-cause hospitalizations | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
Duration of unplanned all-cause hospitalizations | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
Total number of unplanned cardiovascular hospitalizations | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
Duration of unplanned cardiovascular hospitalizations | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
Total number of unplanned hospitalizations related to atrial fibrillation | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
Duration of unplanned hospitalizations related to atrial fibrillation | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
Recurrent unplanned cardiovascular hospitalizations | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
Costs and cost-effectiveness | baseline, 1 year, 2 years, 3 years
  Costs, Quality Adjusted Life Years (QALYs) and Cost-effectiveness (Incremental Cost-Effectiveness Ratio - ICER)
Implementation of care | Follow up with minimum of 1 year and a maximum of 5 years and 10 months
  The extent to which the comprehensive cardiovascular treatment is in accordance with the most recent ESC guidelines Management of Atrial Fibrillation, the HF guidelines of acute and chronic heart failure and the CVD prevention guidelines
Patient Quality of life | Baseline, 1 year, 2 years, 3 years
  General health-related QoL is measured by using the SF-36
Patient Quality of life | Baseline, 1 year, 2 years, 3 years
  Patient's perception of severity of arrhythmia-related symptoms is measured by using the AFSS
Anxiety and/ or depression | Baseline, 1 year, 2 years, 3 years
  HADS-NL
Knowledge of AF | Baseline, 1 year, 2 years, 3 years
  Netherlands Knowledge Scale on AF
Compliance to medication | Baseline, 1 year, 2 years, 3 years
  MMAS
Compliance to medication | Baseline, 1 year, 2 years, 3 years
  To measure the level of activation of a specific individual the PAM-13 Dutch is used

CONTACTS AND LOCATIONS:
Overall Officials: H.J.G.M. Crijns, prof. dr., Principal Investigator — Maastricht University Medical Center; I.C. Van Gelder, prof. dr., Principal Investigator — University Medical Center Groningen; R.G. Tieleman, dr., Principal Investigator — Martini Ziekenhuis
Locations (8):
- Netherlands (8):
  - Martini Ziekenhuis, Groningen
  - UMCG, Groningen
  - Spaarne Gasthuis, Haarlem
  - Medisch Centrum Leeuwarden, Leeuwarden
  - MUMC+, Maastricht
  - Canisius Wilhelmina Ziekenhuis Nijmegen, Nijmegen
  - Zaans Medisch Centrum, Zaandam
  - Isala, Zwolle

REFERENCES:
- [Derived] Wijtvliet EPJP, Tieleman RG, van Gelder IC, Pluymaekers NAHA, Rienstra M, Folkeringa RJ, Bronzwaer P, Elvan A, Elders J, Tukkie R, Luermans JGLM, Van Asselt ADIT, Van Kuijk SMJ, Tijssen JG, Crijns HJGM; RACE 4 Investigators. Nurse-led vs. usual-care for atrial fibrillation. Eur Heart J. 2020 Feb 1;41(5):634-641. doi: 10.1093/eurheartj/ehz666. PMID 31544925